CLINICAL TRIAL: NCT04004637
Title: CD7 CAR-T Cells for Patients With Relapse/Refractory CD7+ NK/T Cell Lymphoma ,T-lymphoblastic Lymphoma and Acute Lymphocytic Leukemia
Brief Title: CD7 CAR-T Cells for Patients With R/R CD7+ NK/T Cell Lymphoma,T-lymphoblastic Lymphoma and Acute Lymphocytic Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-CART-007-001
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: T-lymphoblastic Lymphoma; NK/T Cell Lymphoma; Acute Lymphocytic Leukemia
Keywords: NK/T cell lymphoma; T-lymphoblastic lymphoma; Acute Lymphocytic Leukemia
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Extranodal NK-T-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD7 CAR-T cells Infusion (Experimental)
  Interventions: Drug: CD7 CAR-T cells infusion

INTERVENTIONS:
Drug: CD7 CAR-T cells infusion — Biological: CD7 CAR-T cells infusion. Pretreatment: patients enrolled in this study will receive cyclophosphamide or fludarabine plus cyclophosphamide. CD7 CAR-T cells infusion are allowed within 2 weeks after treatment.
  CD7 CAR-T cells infusion: 30-60 minutes before infusion, H1 anti-histamine agents are applied (acetaminophen 30mg,po.; promethazine 25mg,i.v. ; diphenhydramine 0.5-1mg/kg, no more than 50mg.). Non-physiological doses of corticosteroids are not applied for patients during treatment or recovery unless a life-threatening emergency occurs. CD7 CAR-T cells are infused into patients for one or two times, the number of infused CD7 CAR-T cells are 0.5-5×10^6/kg.

SUMMARY:
This study is designed to explore the safety and efficacy of CD7 CAR-T Cells for patients with relapse/refractory CD7+ NK/T cell lymphoma ,T-lymphoblastic lymphoma and Acute Lymphocytic Leukemia. And to evaluate the pharmacokinetics of CD7 CAR-T cells in patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 7 to 70 years.

  2. The expected survival period is more than 12 weeks.

  3. ECOG: 0-2.

  4. Male and female subjects with CD7+ NK/T cell lymphoma ,T-lymphoblastic lymphoma and Acute Lymphocytic Leukemia in patients with no available curative treatment options will be enrolled:
  1. Not achieved PR after the standard first-line treatment for at least 4 courses.
  2. Relapse or progression after standardized treatment.
  3. Patients With NK/T Cell Lymphoma or T-lymphoblastic Lymphoma need to have at least 1 tumor lesions can be evaluated.

  5. Cardiac left ventricle ejection fraction ≥40%.

  6. Serum creatinine≤1.5 ULN; oxygen saturation of blood >91%.

  7. Total bilirubin≤1.5×ULN; Serum ALT and AST≤2.5 ULN.

  8. Able to understand this study and have signed informed consent.

Exclusion Criteria:

* 1. Patients with graft-versus-host disease (GVHD) or who need to use immunosuppressive drugs.

  2. Patients with malignant tumors other than NK/T cell lymphoma , T-lymphoblastic lymphoma and Acute Lymphocytic Leukemia within 5 years prior to screening, in addition to adequately treated cervical carcinoma in situ, basal or squamous cell skin cancer, local prostate after radical surgery, breast ductal carcinoma in situ after cancer and radical surgery.

  3. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer detection is not within the normal range; hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C Viral (HCV) RNA positive; human immunodeficiency virus (HIV) antibody positive; cytomegalovirus (CMV) DNA positive; syphilis positive.

  4. Severe heart disease: including but not limited to unstable angina pectoris, myocardial infarction (within 6 months prior to screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ III), severe arrhythmia.

  5. Unstable systemic diseases judged by investigator, including but not limited to severe liver, kidney or metabolic diseases needing medical treatment.

  6. Active or uncontrollable infections (except for mild genitourinary infections and upper respiratory tract infections) that require systemic treatment within 7 days prior to screening; 7. Women who are pregnant or breastfeeding, female subject who plans to have a pregnancy within 1 year after cell infusion, and male subject who plans to have a pregnancy within 1 year after cell infusion.

  8. Subject who have received CAR-T treatment or other genetically modified cell therapy before screening; 9. Subjects who are receiving systemic steroid therapy within 7 days prior to screening or who require long-term systemic steroid therapy judged by investigator (except for inhaled or topical use); 10. Participated in other clinical studies within 3 months prior to screening. 11. Patients with active CNS involvement by malignancy. 12. Not suitable for cell preparation. 13. Researchers consider it inappropriate to participate in the trial.

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-08-25 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Identification of the dose limiting toxicity (DLT) | Time Frame: 4 weeks after CAR T cell infusion
  Toxicity will be assessed according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) scale, version 5 and the number of patients experiencing DLT will be evaluated.

SECONDARY OUTCOMES:
In vivo persistence/expansion of infused CAR T cell | Up to 2 years
  Detection of infused CAR T cell in the peripheral blood.
Determine the effects of CART-CD7 infusion on T cells and CD7 expression in vivo. | Up to 2 years
Overall Response Rate (ORR) | 4 weeks after CAR T cell infusion
Overall Survival | Up to 2 years
Disease-free survival | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang M, Chen D, Fu X, Meng H, Nan F, Sun Z, Yu H, Zhang L, Li L, Li X, Wang X, Wang M, You F, Li Z, Chang Y, Zhou Z, Yan J, Li J, Wu X, Wang Y, Wang Y, Xiang S, Chen Y, Pan G, Xu H, Zhang B, Yang L. Autologous Nanobody-Derived Fratricide-Resistant CD7-CAR T-cell Therapy for Patients with Relapsed and Refractory T-cell Acute Lymphoblastic Leukemia/Lymphoma. Clin Cancer Res. 2022 Jul 1;28(13):2830-2843. doi: 10.1158/1078-0432.CCR-21-4097. PMID 35435984